CLINICAL TRIAL: NCT04451434
Title: A Phase 1 Study to Determine the Safety, Tolerability, and Pharmacokinetics of Danicopan After Administration as an Oral Tablet in the Fed and Fasted States in Participants of Japanese Descent
Brief Title: Study of Danicopan in Participants of Japanese Descent
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ALXN2040-HV-101
Record Dates: First submitted 2020-06-19; First posted 2020-06-30 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: Factor D inhibitor; Complement; Danicopan; Pharmacokinetics; Japanese; Food
MeSH Terms: interventions — danicopan

STUDY DESIGN:
Intervention Model Description: Three-way crossover
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Danicopan 200 mg Fasted (Experimental): Fasting participants will receive a single dose of 200 mg danicopan.
  Interventions: Drug: Danicopan
- Danicopan 200 mg Fed (Experimental): Fed participants will receive a single dose of 200 mg danicopan.
  Interventions: Drug: Danicopan
- Danicopan 400 mg Fed (Experimental): Fed participants will receive a single dose of 400 mg danicopan.
  Interventions: Drug: Danicopan

INTERVENTIONS:
Drug: Danicopan — Oral tablet
  Other Names: ALXN2040; ACH-0144471

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of danicopan after a single-dose oral administration under fed and fasting conditions to participants of Japanese descent.

DETAILED DESCRIPTION:
This will be an open-label, randomized, single-dose, 3-period, 3-treatment crossover study in participants of Japanese descent.

On Day 1 of each period, participants will receive a single oral dose of 200 milligrams (mg) danicopan under fasting conditions, 200 mg danicopan under fed conditions, or 400 mg danicopan under fed conditions. Participants will receive each treatment once, according to the randomization schedule. There will be a washout period of at least 7 days between each dose of study intervention.

Safety will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are of Japanese descent defined as:

   * First generation (born to 2 Japanese parents and 4 Japanese grandparents)
   * Born in Japan, and not have lived outside Japan for greater than 10 years
   * Lifestyle, including diet, must not have significantly changed since leaving Japan
2. No clinically significant history or presence of electrocardiogram findings as judged by the Investigator at screening and prior to the first dose of study intervention in Period 1.
3. Body mass index in the range of 18.0 to 32.0 kilograms (kg)/meters squared, inclusive, with a minimum body weight of 50.0 kg at screening.

Exclusion Criteria:

1. Evidence of any clinically significant deviation from normal in clinical laboratory evaluations, as determined by the Investigator or designee.
2. History of any medical or psychiatric condition or disease that, in the opinion of the Investigator or designee, might limit the participant's ability to complete or participate in this clinical study, confound the results of the study, or pose an additional risk to the participant by their participation in the study.
3. History or presence of clinically significant hypersensitivity or idiosyncratic reaction to the study interventions or related compounds or commonly used antibacterial agents.
4. History of meningococcal infection, or a first-degree relative with a history of meningococcal infection.
5. History of febrile illness, or other evidence of infection, within 14 days prior to the first dose of study intervention.
6. Any major surgery within 4 weeks of the first dose of study intervention.
7. Diagnosis or history of Gilbert's syndrome, in the opinion of the Investigator or designee.
8. Unable to refrain from or anticipates the use of any drug.
9. Receipt of a vaccine within 30 days prior to the first dose of study intervention.
10. Receipt of blood products within 6 months prior to the first dose of study intervention.
11. Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives (if known) or 30 days prior to the first dose of study intervention, whichever is longer.
12. Seated blood pressure is less than 90/40 millimeters of mercury (mmHg) or greater than 140/90 mmHg at screening.
13. Participants who test positive for human immunodeficiency virus, hepatitis B virus, and/or hepatitis C virus.
14. Current tobacco users and smokers or a positive cotinine test at screening.
15. Donation of whole blood from 3 months prior to the first dose of study intervention, or of plasma from 30 days prior to the first dose of study intervention.
16. Positive drugs of abuse screen at screening or Day -1 of Period 1.
17. Positive results for alcohol screen at screening or Day -1 of Period 1.
18. Is a female with a positive pregnancy test at screening or Day -1 of Period 1 or who is lactating, or who plan to become pregnant (within 5 months of screening).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Number Of Participants With Treatment-Emergent Adverse Events | Day 1 (after first dose) through safety follow-up (10 +/- 2 days after last dose)
Area Under The Concentration Versus Time Curve (AUC) Of Danicopan In Both Fed And Fasted States | up to 72 hours postdose
Maximum Observed Concentration (Cmax) Of Danicopan In Both Fed And Fasted States | up to 72 hours postdose
Time To Maximum Observed Concentration (Tmax) Of Danicopan In Both Fed And Fasted States | up to 72 hours postdose
Dose Proportionality Of Danicopan In Fed State Assessed by AUC | up to 72 hours postdose
Dose Proportionality Of Danicopan In Fed State Assessed by Cmax | up to 72 hours postdose

SECONDARY OUTCOMES:
Activity Of Danicopan As Measured By Alternative Pathway Wieslab Assay | up to 72 hours postdose
  Blood samples will be collected for measurement of danicopan activity.
Complement Factor B Fraction b Levels | up to 72 hours postdose
  Blood samples will be collected for measurement of complement factor B fraction b levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Study Site, Brisbane, Australia

IPD SHARING:
Plan to Share IPD: No